CLINICAL TRIAL: NCT03553563
Title: An Open Label, Parallel Group, Multi-centre, Phase III Study to Assess the Efficacy and Safety of D961H for the Maintenance Therapy Following Initial Treatment in Japanese Paediatric Patients With Reflux Esophagitis and for the Prevention of Recurrence of Gastric Ulcer or Duodenal Ulcer in Japanese Paediatric Patients Treated With Non-steroidal Anti-inflammatory Drugs or Low-dose Aspirin
Brief Title: A Study of Esomeplazole (D961H) in Japanese Paediatric Patients With Reflux Esophagitis, Gastric Ulcer or Duodenal Ulcer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D961WC00001; 2018-000213-20 (EudraCT Number)
Record Dates: First submitted 2018-04-05; First posted 2018-06-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Reflux Esophagitis; Gastric Ulcer; Duodenal Ulcer
Keywords: D961H; paediatric; reflux esophagitis; gastric ulcer
MeSH Terms: conditions — Esophagitis, Peptic; Stomach Ulcer; Duodenal Ulcer | interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: An open label, parallel four group, multi-centre, phase III study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group1 (Experimental): Initial healing phase (8 weeks), D961H 10 mg once-daily; Maintenance phase (24 or 44 weeks), D961H 10 mg once-daily
  Interventions: Drug: D961H capsule 10mg; Drug: D961H sachet 10mg
- Group2 (Experimental): Initial healing phase (8 weeks), D961H 20 mg once-daily; Maintenance phase (24 or 44 weeks) starts with D961H 10 mg once-daily and may be increased to 20 mg once-daily based on investigator's discretion
  Interventions: Drug: D961H capsule 10mg; Drug: D961H sachet 10mg
- Group3 (Experimental): D961H 10 mg once-daily (32 or 52 weeks)
  Interventions: Drug: D961H capsule 10mg; Drug: D961H sachet 10mg
- Group4 (Experimental): D961H starts with 10 mg once-daily, and may be increased to 20 mg once-daily based on investigator's discretion (32 or 52 weeks)
  Interventions: Drug: D961H capsule 10mg; Drug: D961H sachet 10mg

INTERVENTIONS:
Drug: D961H capsule 10mg — All Groups can select either capsule or sachet during the study.
  Other Names: esomeprazole
Drug: D961H sachet 10mg — All Groups can select either capsule or sachet during the study.
  Other Names: esomeprazole

SUMMARY:
This is an open label, parallel group, multi-centre, phase III study to assess the safety and efficacy of D961H in maintenance therapy following initial healing therapy in Japanese paediatric patients with reflux esophagitis, and to assess the safety and efficacy of D961H in Japanese paediatric patients treated with long term non-steroidal anti-inflammatory drugs or low-dose aspirin therapy who have a documented medical history of gastric ulcer or duodenal ulcer diagnosis.

Doses of D961H in this study is set for the 2 groups (weight more than equal 10 kg to less than 20 kg and weight more than equal 20 kg) in the maintenance therapy for healed reflux esophagitis group and the prevention of gastric ulcer or duodenal ulcer recurrence by non-steroidal anti-inflammatory drugs or low-dose aspirin therapy group, Primary endpoints are evaluated at week 32. Further, this study is designed to evaluate the long term efficacy and safety of D961H for a maximum of 52 weeks, in consideration of the medical needs for long term proton pump inhibitor treatment. Patient can continue study treatment up to 52 weeks, if they want

DETAILED DESCRIPTION:
Subjects are allocated to four groups based on their disease and weight.

Number of Subjects

Maintenance therapy for healed reflux esophagitis study part:

* Group1:aged 1 to 14 years (weight more than equal 10 kg to less than 20 kg ), Maintenance phase, n=5 to 10
* Group2:aged 1 to 14 years (weight more than equal 20 kg), Maintenance phase, n=10 to 20

Prevention of gastric ulcer or duodenal ulcer recurrence associated with long term non-steroidal anti-inflammatory drugs or low-dose aspirin therapy study part:

* Group3:aged 1 to 14 years (weight more than equal 10 kg to less than 20 kg), n=5 to 10 at Week 0
* Group4:aged 1 to 14 years (weight more than equal 20 kg), n=10 to 20 at Week 0

All subjects have a D961H administration for 32 or 52 weeks. all esophagogastroduodenoscopy findings are reviewed by central evaluation committee and study is conducted based on the judgement of central evaluation committee.

Data are entered in electric data capture system at study site by site staffs and all data are verified with source data by site monitors during the study.

Analyses will be performed by AstraZeneca or its representatives. A comprehensive statistical analysis plan will be developed and finalised before database lock and will describe the subject populations to be included in the analyses, and procedures for accounting for missing, unused, and spurious data. This section is a summary of the planned statistical analyses of the primary and secondary endpoints. Any deviations from this plan will be reported in the clinical study report.

Efficacy analyses are intended for Efficacy Analysis Set. ・Efficacy Analysis Set:All subjects who take at least 1 dose of the investigational product and have at least 1 efficacy datum assessment during the maintenance/prevention therapy period, and who have no important protocol deviation.

All safety analyses are performed on the Safety Analysis Set.

・Safety Analysis Set:All subjects who take at least 1 dose of the investigational product and have any post-treatment assessment.

Frequency and incidence rate of adverse events (AEs), serious adverse events (SAEs), discontinuation of investigational product due to adverse events (DAEs) and other significant adverse events (OAEs) will be presented by MedDRA System Organ Class (SOC) and Preferred Term (PT) for each group. In addition, summaries of AEs will be further broken down by maximum intensity and relationship to the investigational product as assigned by investigators

ELIGIBILITY:
Inclusion Criteria:

For healed reflux esophagitis study

* Endoscopically verified reflux esophagitis, Grade A or higher according to the Los Angels classification as judged by central evaluation committee.

For prevention of gastric ulcer or duodenal ulcer recurrence study

* Patients with documented medical history of gastric ulser or duodenal ulser diagnosis based on upper gastrointestinal symptoms, fecal occult blood, esophagogastroduodenoscopy findings, etc.

Exclusion Criteria:

* Patients less than 10 kg in weight.
* Use of any other investigational compounds or participations in another clinical trial within 4 weeks prior to the enrolment.
* Significant clinical illness within 4 weeks prior to the informed consent
* Previous total gastrectomy.
* Presence of hepatic diseases or other conditions that could interfere with evaluation of the study as judged by investigators. etc.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Presence/absence of reflux esophagitis relapse | 8 to 32 weeks
  Maintenance therapy for healed reflux esophagitis study part:
  Presence/absence of reflux esophagitis relapse from 8 to 32 weeks for all subjects by assessment of the composite endpoint (reflux esophagitis -related symptoms or optional esophagogastroduodenoscopy findings) during the maintenance therapy.
Adverse events during reflux esophagitis maintenance therapy | 8 to 32 weeks
  Maintenance therapy for healed reflux esophagitis study part:
  Safety from 8 to 32 weeks for all subjects.
Presence/absence of gastric ulcer or duodenal ulcer recurrence | 0 to 32 weeks
  Prevention of gastric ulcer or duodenal ulcer recurrence associated with long term non-steroidal anti-inflammatory drugs or low-dose aspirin therapy study part:
  Presence/absence of gastric ulcer or duodenal ulcer recurrence from 0 to 32 weeks for all subjects by assessment of the composite endpoint (gastric ulcer or duodenal ulcer-related symptoms or optional esophagogastroduodenoscopy findings) during the prevention therapy.
Adverse events during gastric ulcer or duodenal ulcer recurrence prevention therapy | 0 to 32 weeks
  Prevention of gastric ulcer or duodenal ulcer recurrence associated with long term non-steroidal anti-inflammatory drugs or low-dose aspirin therapy study part:
  Safety from 0 to 32 weeks for all subjects.

SECONDARY OUTCOMES:
Presence/absence of reflux esophagitis relapse | 8 to 52 weeks
  Presence/absence of reflux esophagitis relapse from 8 to 52 weeks for subjects who continued the study treatment after Week 32 by assessment of the composite endpoint (reflux esophagitis-related symptoms or optional esophagogastroduodenoscopy findings) during the maintenance therapy.
Adverse events during reflux esophagitis maintenance therapy | 8 to 52 weeks
  Maintenance therapy for healed reflux esophagitis study part:
  Safety from 8 to 52 weeks for subjects who continued the study treatment after Week 32.
Presence/absence of gastric ulcer or duodenal ulcer recurrence | 0 to 52 weeks
  Presence/absence of gastric ulcer or duodenal ulcer recurrence from 0 to 52 weeks for subjects who continued the study treatment after Week 32 by assessment of the composite endpoint (gastric ulcer or duodenal ulcer-related symptoms or optional esophagogastroduodenoscopy findings) during the prevention therapy.
Adverse events during gastric ulcer or duodenal ulcer recurrence prevention therapy | 0 to 52 weeks
  Prevention of gastric ulcer or duodenal ulcer recurrence associated with long term non-steroidal anti-inflammatory drugs or low-dose aspirin therapy study part:
  Safety from 0 to 52 weeks for subjects who continued the study treatment after Week 32.

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Shimizu, M.D., Ph.D., Study Chair — Juntendo University Graduate School of Medicine
Locations (15):
- Japan (15):
  - Research Site, Bunkyō City
  - Research Site, Fuji-shi
  - Research Site, Izumi-shi
  - Research Site, Kagoshima
  - Research Site, Kanazawa
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Matsumoto-shi
  - Research Site, Okayama
  - Research Site, Saitama-shi
  - Research Site, Sakaishi
  - Research Site, Setagaya-ku
  - Research Site, Shinjuku-ku
  - Research Site, Takatsuki-shi
  - Research Site, Yokohama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home